CLINICAL TRIAL: NCT03760094
Title: Role of Color Doppler Ultrasound in Differentiation Between Benign and Malignant Lymphadenopathy
Brief Title: Role of Color Doppler Ultrasound in Lymphadenopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Gergis Naeem, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Color Doppler Ultrasound
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Lymph Node Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): patients with lymphadenopathy
  Interventions: Device: Colour Doppler

INTERVENTIONS:
Device: Colour Doppler — evaluation of lymph nodes by Doppler

SUMMARY:
Lymphadenopathy is defined as an abnormality in the size or character of lymph nodes caused by the invasion or propagation of either inflammatory or neoplastic cells into the nodes Accurate lymph node characterization is important for a wide number of clinical situations, including prognosis, prediction, selecting and monitoring treatment, beyond the diagnosis itself (cancer, lymphoma, or inflammatory nodes)

DETAILED DESCRIPTION:
Various ultrasound criteria that can help in differentiation of benign and malignant lymph nodes have been well described in literature. On Gray scale ultrasound imaging, the benign enlarged lymph nodes are hypoechoic, oval shaped with smooth border and echogenic hilum. On the other hand, the malignant lymph nodes are round with short to long axis ratio >0.5 and show loss of echogenic hilum, while the Color and Power Doppler features documented for the diagnosis of malignant lymph nodes are peripheral and mixed vascularity, with resistive index (RI) more than 0.8, and pulsatility index (PI) more than 1.5 Although Color Doppler ultrasound improves diagnostic accuracy and plays an important adjuvant role to Gray scale ultrasound in differentiating benign from malignant lymph nodes as it adds to the diagnostic confidence of predicting malignancy in enlarged lymph nodes, and also is useful if Gray scale ultrasound findings are equivocal. However, it can neither replace histopathology nor can eliminate the need for biopsy

ELIGIBILITY:
Inclusion Criteria:

* clinically enlarged lymph nodes

Exclusion Criteria:

* previous medical treatment or radiotherapy
* previous biopsy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with benign lymphadenopathy | one year
  comparison with the biopsy result